CLINICAL TRIAL: NCT00249171
Title: Comparison of Oral Risperdal in Combination With Oral Lorazepam vs Standard Care Including Initial Conventional Neuroleptic IM Treatment, in Acute Schizophrenic Patients
Brief Title: A Study of Risperidone in Combination With Lorazepam Compared With Standard Therapy for Emergency Treatment of Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003175
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia; Psychotic Disorders; Emergency Treatment
Keywords: acute schizophrenia; psychosis; risperidone; lorazepam, antipsychotic agents; emergency treatment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of the study is to show that risperidone (an antipsychotic medication) combined with lorazepam (an anti-anxiety medication) is more effective than conventional therapy administered by intramuscular injection for emergency treatment of patients with schizophrenia.

DETAILED DESCRIPTION:
Patients with acute schizophrenia are often anxious and uncertain because of the psychotic symptoms they are experiencing. These patients are in need of rapid help and symptom relief. Risperidone, a widely used antipsychotic medication, is effective against positive and negative symptoms of schizophrenia, has a rapid onset of action, a low incidence of extrapyramidal symptoms, and, in general, mild adverse events. This is an open-label trial of 2 mg dose of an oral formulation of risperidone in combination with 2 to 2.5 mg of oral lorazepam compared with standard care, which consists of a conventional neuroleptic drug administered via an intramuscular injection, with or without lorazepam. Patients requiring emergency care are offered a choice of these two therapies and are monitored for 24 hours after initial treatment. Optional follow up may be performed after 2, 3, and 7 days. The primary measure of effectiveness is the success of the treatment 2 hours after the drug is administered, as indicated by the patient being asleep or by showing improvement on the Clinical Global Impression (CGI) Improvement subscale. Additional effectiveness assessments include an evaluation of hostility and agitation, as assessed by Brief Psychiatric Rating Scale (BPRS), the degree of sedation, and the ability of the patient to interact with the physician at 1, 2, and 24 hours after the start of treatment. Safety assessments include the incidence of adverse events throughout the treatment and follow up periods. The study hypothesis is that oral risperidone combined with lorazepam is more effective than therapy with conventional neuroleptic intramuscular agents, with or without lorazepam, for emergency treatment of patients with schizophrenia. Single, oral 2 mg dose of risperidone and a single, oral 2 to 2.5 mg dose of lorazepam; further dosing during the 24 hour period at investigator's discretion. Comparator drug of choice (with or without lorazepam) administered intramuscularly according to product labeling.

ELIGIBILITY:
Inclusion Criteria:

* Psychotic patients with schizophrenia who require rapid intervention
* experiencing symptoms of a psychotic disorder
* capable of choosing to be treated

Exclusion Criteria:

* Patients with a known hypersensitivity to the study drugs
* have participated in an investigational drug trial within 30 days of study initiation
* known to be unresponsive to treatment with risperidone or the comparator drug
* known to have benzodiazepine dependence (addiction to this class of anti-anxiety drugs)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2001-06; Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Treatment success, 2 hours after drug administration, indicated by patient being asleep or by improvement on Clinical Global Improvement (CGI) scale.

SECONDARY OUTCOMES:
Hostility and agitation (as assessed by BPRS), degree of sedation, and ability to interact with physician at 0, 1, 2, and 24 hours; Clinical Global Impression (CGI) - Improvement subscale at 1 and 24 hours; adverse events throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Lejeune J, Larmo I, Chrzanowski W, Witte R, Karavatos A, Schreiner A, Lex A, Medori R. Oral risperidone plus oral lorazepam versus standard care with intramuscular conventional neuroleptics in the initial phase of treating individuals with acute psychosis. Int Clin Psychopharmacol. 2004 Sep;19(5):259-69. doi: 10.1097/01.yic.0000138820.78121.0e. PMID 15289699